CLINICAL TRIAL: NCT00847522
Title: Fluorescein for Lymphatic Mapping and Sentinel Lymph Node Biopsy in Patients With Stage I and II Malignant Melanoma
Brief Title: Fluorescein for Lymphatic Mapping and Sentinel Lymph Node (SLN) Biopsy in Patients With Stage I and II Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCI26818
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: melanoma; skin cancer; lymph node; sentinel lymph node; malignant melanoma; mapping
MeSH Terms: conditions — Neoplasms; Melanoma; Skin Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: 10 patients were enrolled in the Phase 1 portion of the trial. 80 patients were enrolled in the Phase 2 portion of the trial. 90 patients were enrolled total for the Phase 1 and 2 portions. Results are reported for the 80 patients on the Phase 2 portion.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Fluorescein

INTERVENTIONS:
Drug: Fluorescein — Fluorescein is an orange-red powdered compound, designated by the formula C20H12O5, which exhibits intense greenish-yellow fluorescence in alkaline solution. It has been used extensively in surgery and medicine for decades for diagnostic purposes. Topical fluorescein is routinely used in ophthalmology to assess corneal lesions. Intravenous fluorescein is used in vascular surgery to measure vascular perfusion and in skin and melanoma surgery to assess the viability of skin flaps.
  Other Names: Fluorescite®

SUMMARY:
The purpose of this research study is to use two different drugs to find where melanoma might spread and to remove these tissues. We believe that tumor cells from the melanoma first move through the lymphatic system (a system of clear fluid that moves around the body and carries white blood cells, much like the blood system) to a lymph node in an orderly way. If we can identify the first lymph nodes to receive a tumor cell, this can be removed and examined. We currently use one drug, called "technetium-99m sulfur colloid" which can detect about 90% of the first lymph nodes that the tumor cells would move to. Technetium-99m is a radioactive compound and can be detected through the skin by a special instrument that reads radioactivity. As part of this research, we would like to use a second drug called "fluorescein" (Fluorescite®) to see if it will identify the same lymph nodes or additional ones and examine these. This drug is fluorescent and can be detected even through the skin using a blue light. This drug is approved by the Federal Drug Administration (FDA) to for injection in the vein as a diagnostic aid and has been safely used in people for many years. In this study, we will be injecting it under the skin, which is a different use from how it is currently approved by the FDA. In the past another drug has been used, called "isosulfan blue" (Lymphazurin®), but availability of this drug is currently limited, and it has higher risks associated with it.

This study is being conducted by Dr. Robert Andtbacka, Dr. Dirk Noyes, Dr. James McGreevy and at University of Utah. This study is a Phase I/II and is done to find out if the drug can be used safely when given under the skin and if it will work for this purpose.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary goal of this study is to evaluate the ability of intradermal fluorescein to detect sentinel lymph nodes (SLNs) in patients with stage I and stage II melanoma.

Primary Objectives To determine the co-localization between fluorescein and technetium-99m labeled sulfur colloid in SLNs.

Secondary Objectives

1. To evaluate the toxicity and safety of intradermal fluorescein injections.

The management of regional lymph nodes in patients with clinically localized primary melanomas has been controversial. An elective lymph node dissection at the time of removal of the primary melanoma has been favored by many. The proponents of elective lymph node dissection has based their opinion of the hypothesis that melanoma spreads in an orderly fashion from the primary site to regional lymph nodes and then systemically. Thus early removal of lymph node tumor deposits may prevent subsequent systemic dissemination.1-7 Four prospective randomized trials of elective lymphadenectomy have tested this hypothesis.8-11 In all of these trials, elective lymphadenectomy did not result in a significant survival benefit. In one of the trials8, a subgroup analysis indicated that elective lymphadenectomy may benefit patients younger than 60 years of age, especially those with nonulcerated primary melanomas and melanomas between 1-2mm in thickness. Based on these results, elective lymphadenectomy for patients with stage I and II melanoma is not advocated and this has resulted in a more selective evaluation of the regional lymph nodes and development of the sentinel lymph node biopsy (SLNB) technique.

The sentinel lymph node (SLN) concept is based on the hypothesis that tumor cells from primary melanomas metastasizes through the lymphatic system to regional lymph nodes in an orderly fashion and that mapping of the lymphatic system can identify the first or "sentinel" lymph node to receive metastatic tumor cells. This sentinel lymph node will become involved with metastasis before any other node in the regional lymph node basis and if involved will reflect the pathologic status of the entire regional nodal basin. Morton et al.12 were the first to evaluate the SLN concept in patients with stage I melanoma. In this study of 237 lymph node basins in 233 patients, the SLN was identified 82% of the time and it predicted the pathologic status of the nodal basin in 99% of cases. Since this preliminary study, substantial progress has been made improving and standardizing the techniques for lymphatic mapping and SLNB.

Use of a vital blue dye such as 1% isosulfan blue (Lymphazurin®) has been part of the lymphatic mapping and SLNB since its introduction. At the time of operation, 3-5 ml of the vital blue dye is injected intradermally around the intact primary melanoma or the tumor biopsy site. The dye rapidly diffuses into the lymphatic system and is carried by afferent lymphatic trunks to the SLN. An incision is made over the draining nodal basin and the blue afferent lymphatic channels are followed to the first draining lymph node(s), the sentinel lymph nodes. With the use of a vital blue dye, the SLN can be identified in approximately 87% of cases.13 This leaves 13% of patients unable to benefit from a SLN evaluation. Gershenwald et al. demonstrated that SLN identification improved from 87% to 99% when technetium-99m labeled sulfur colloid was combined with the vital blue dye. 13 To increase the detection rate of SLNs, two additional techniques are commonly used: a) pre-operative lymphoscintigraphy using a technetium-99m labeled sulfur colloid or human albumin radiotracer 14, 15 to better delineate the lymphatic drainage and identify multiple drainage basins and b) intraoperative use of a handheld gamma probe to better localize the SLN. Currently, using the vital blue dye technique in combination with a radiotracer identifies the SLN in up to 99% of cases.13, 16, 17 Based on these findings, most clinicians now recommend using a combined modality approach which is considered the "gold standard" for SLN localization in patients with primary melanoma. Although the technetium-99m labeled sulfur colloid adds a greater detection ability, formal studies have not been reported using this alone. Informal observation finds that one can pick up radioactivity in nodes which are not blue more often than one picks up blue nodes that are not radioactive, but again the ideal situation is to be able to use two tracers at once.

Although 1% isosulfan vital blue dye increases the detection of SLNs when combined with a radiotracer, it has several drawbacks. First, the dye can diffuse throughout the operative wounds making dissection and SLN identification difficult. This is especially concerning if the afferent lymphatic channels are cut. Second, 1% isosulfan blue dye has been associated with an anaphylactoid reaction or a life threatening anaphylactic shock in 0.1 - 2% of patients undergoing lymphatic mapping and SLNB.18-23 Third, a recent shortage in 1% isosulfan blue has resulted in a decreased access to the compound for patients and clinicians. Thus, there is a great need to develop new lymphatic mapping and SLN identification techniques.

Fluorescein is an orange-red powdered compound, designated by the formula C20H12O5, which exhibits intense greenish-yellow fluorescence in alkaline solution. It has been used extensively in surgery and medicine for decades for diagnostic purposes. Topical fluorescein is routinely used in ophthalmology to assess corneal lesions.24 Intravenous fluorescein is used in vascular surgery to measure vascular perfusion25 and in skin and melanoma surgery to assess the viability of skin flaps.26, 27 Intradermal fluorescein injections have been used to identify pedal lymphatics to facilitate lymphangiography.28 This study was designed to look at both the safety and efficacy of using 10% fluorescein mixed 1:1 with 1% lidocaine hydrochloride. Cooper et al. reported on intradermal injection of fluorescein in 1,047 patients without adverse reactions.28 In this study, "not a single immunologic reaction was identified. In two patients, local skin sloughing occurred at the injection site due to inadvertent administration of a 3;1 fluorescein-lidocaine mixture rather than the prescribed 1:1 ratio". Dan et al.29 used intramural bowel injection of fluorescein in 120 patients with colon cancer to map the lymphatics in patients with colon cancer. Fluorescein was able to identify the sentinel lymph node in 97% of patients and none of the 120 patients suffered any adverse reactions. We have previously shown that Cy5-cobolamine bioconjugate injected intradermally into the hind limb of pigs is able to identify inguinal sentinel lymph nodes.30 More recently, we have also determined that fluorescein injected intradermally into the limb of pigs is also able to identify the sentinel lymph node. Additionally, when 1% isosulfan blue is injected in the same location as fluorescein, the two detection techniques co-localizes in the afferent lymphatics and the sentinel lymph node. The fluorescent signal from fluorescein provides improved detection of the afferent lymphatic and the sentinel lymph node compared to 1% isosulfan blue. Moreover, fluorescein fluorescence is clearly visualized transdermally and enables an improved localization of the sentinel lymph node prior to performing a skin incision. (Andtbacka RH, McGreevy JM, Grissom CB et al. unpublished results). This transdermal fluorescence may enable elimination of the radiotracer in sentinel lymph node detection. Based on these findings we are now proposing a phase I/II clinical trial in melanoma to assess the safety and feasibility of intradermal fluorescein in the detection of SLNs in patients with stage I and stage II melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.
2. Between 18 and 90 years of age.
3. Have a primary melanoma that is cutaneous (including head, neck, trunk, extremity, scalp, palm, sole, subungual skin tissues)
4. Have a primary melanoma meeting one of the following criteria:

   1. Primary melanoma was ≥ 0.75 mm Breslow thickness and Clark level III or
   2. Primary melanoma was Clark level IV/V or
   3. Primary melanoma was ulcerated or
   4. Primary tumor mitotic >1/mm2 or
   5. Primary melanoma was less than 0.75 mm Breslow thickness with one or more poor prognostic features (regression > 75%, vertical growth phase, mitotic Count > 1/mm2, transected deep biopsy margin) or
   6. Have had a prior excision (non-wide local excision) of a melanocytic lesion with development of a primary melanoma in the excision scar or
   7. Have had a wide locale excision within the past 120 days of a primary melanoma as defined in (a-f) above but not yet undergone a SLNB
5. Clinically negative lymph nodes.
6. ECOG performance status 0-1

Exclusion Criteria:

1. Primary melanoma of the eye, mucous membranes or internal viscera.
2. Physical, clinical, radiographic or pathologic evidence of satellite, in-transit, regional or distant metastatic disease.
3. Skin grafts, tissue transfers or flaps that have the potential to alter the lymphatic drainage pattern from the primary melanoma to the lymph node basin.
4. Allergy to radiocolloid or fluorescein.
5. Inability to localize 1-2 SLN drainage basins via lymphatic mapping. (e.g., no basin found which emits gamma-radiation after injection with technecium-99m or more than 2 basins are found which emit gamma-radiation.)
6. Prior completion lymph node dissection or SLNB that may have altered the lymphatic drainage from the primary cutaneous melanoma to a potential lymph node basin.
7. Organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the protocol, or be exacerbated by therapy.
8. Melanoma-related operative procedures not corresponding to criteria described in the protocol.
9. Primary or secondary immune deficiencies or known significant autoimmune disease which would pose a risk to the participant based on the physician's judgment.
10. History of organ transplantation.
11. Pregnant or lactating women.
12. Participation in concurrent experimental protocols or alternative therapies that might confound the analysis of this trial. Adjuvant therapy protocols after recurrence are acceptable.
13. Nonmalignant systemic disease (e.g., cardiovascular, renal, hepatic, etc.) that precludes a patient from being subjected to any of the treatment options or that would prevent prolonged follow-up based on the physician's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Andtbacka, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Phase II study with dose of VST-001 set at 5ml fluorescein sodium 0.01% solution administered intradermally for intraoperative lymphatic mapping in patients with Stage I or II malignant melanoma.
  Fluorescein: Fluorescein is an orange-red powdered compound, designated by the formula C20H12O5, which exhibits intense greenish-yellow fluorescence in alkaline solution. It has been used extensively in surgery and medicine for decades for diagnostic purposes. Topical fluorescein is routinely used in ophthalmology to assess corneal lesions. Intravenous fluorescein is used in vascular surgery to measure vascular perfusion and in skin and melanoma surgery to assess the viability of skin flaps.
Period: Overall Study
Arm/Group | All Patients
Started | 90
Phase I | 10
Phase II | 80
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 90
Age, Continuous [Median (Full Range); unit: years] | 50.5 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Agreement Between the Detection of SLNs
Description: There is compete agreement if there are no SLNs that are either radioactive only or fluorescent only via intradermal fluorescein and technetium-99m labeled sulfur colloid.
Time Frame: 2 days
Population: Total number of patients with at least one SLN was 89
Measure: Number; unit: percentage complete agreement
Arm/Group | All Patients
Number analyzed (Participants) | 89
percentage complete agreement | 69.7

2. Secondary Outcome: Safety Evaluation of Intradermal Fluorescein Injections.
Description: Number of participants that experienced an adverse event
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 90
Participants
  Adverse Event Recorded | 5
  Adverse Events Related to Study Treatment | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: All Adverse Events are reported - none were considered related to the investigational product.
Groups:
- Phase I/II Patients: Fluorescein: Fluorescein is an orange-red powdered compound, designated by the formula C20H12O5, which exhibits intense greenish-yellow fluorescence in alkaline solution. It has been used extensively in surgery and medicine for decades for diagnostic purposes. Topical fluorescein is routinely used in ophthalmology to assess corneal lesions. Intravenous fluorescein is used in vascular surgery to measure vascular perfusion and in skin and melanoma surgery to assess the viability of skin flaps.
Arm/Group | Phase I/II Patients
All-Cause Mortality (participants affected / at risk) | 5/90
Serious Adverse Events (participants affected / at risk) | 1/90
Other Adverse Events (participants affected / at risk) | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II Patients (N=90)
hematoma, scalp pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II Patients (N=90)
wound infection (Infections and infestations) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
neurophathic pain (Nervous system disorders) | 1 (1)
amnesia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes